CLINICAL TRIAL: NCT05842005
Title: Mesh-Reduced Sling For Treating Stress Urinary Incontinence, Efficacy and Durability Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Henry Chill, Principal Investigator, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH22-464
Record Dates: First submitted 2023-04-18; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Stress Urinary Incontinence
Keywords: Mesh-reduced sling; Safety; Efficacy; Treatment
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective case series. Our hypothesis is that the mesh-reduced sling will improve stress urinary incontinence (SUI) symptoms in women with SUI and normal urethral closure pressure at 2 months and 12 months after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mesh-reduced Sling (Experimental): Mesh-reduced sling will improve stress urinary incontinence (SUI) symptoms in women with SUI and normal urethral closure pressure at 2 months and 12 months after surgery.
  Interventions: Device: Mesh-reduced Sling

INTERVENTIONS:
Device: Mesh-reduced Sling — In this proposed study, the investigators aim to evaluate the role of using a ¾ x ⅜ inch cm polypropylene mesh suspended by sutures as a mesh-reduced solution for SUI.

SUMMARY:
The goal of this pilot study is to report the safety and efficacy of a suture-suspended mesh-reduced sling for treating stress urinary incontinence (SUI) in women.

The main question[s] it aims to answer are:

* investigate the efficacy of this mesh-reduced suture-based surgical technique for improving SUI symptoms
* investigate the efficacy of this mesh-reduced suture-based surgical technique on key urethral support defects observed with 3D ultrasound Participants will consent to participate following which they will complete pre-operative assessments according to our routine clinical pathway. The participant will then undergo surgery and will be followed up to 12 months post-operatively via symptom assessment and pelvic exam.

DETAILED DESCRIPTION:
Women presenting to our tertiary urogynecology clinic with stress urinary incontinence symptoms based on their answers to PFDI-20 questionnaire and deciding to proceed with surgical treatment of SUI will be invited to participate in this study. Baseline screening will include our standard clinical pathway, which includes symptom review and standard questionnaires, standard vaginal and, urodynamic study and 3D pelvic floor ultrasound. If clinical and ultrasound imaging findings are consistent with SUI in setting of normal urethral closure pressure but lack of urethral support that is state of the art indication for mid-urethral sling procedure, patients will be offered this mesh-reduced mini-sling mesh-reduced sling for treating their condition.

For patients expressing interest, the study procedures and consent will be reviewed during this office visit. Consent will be signed at the following pre-op visit. This study will involve no additional pre-operative tests or questionnaires, beyond our routine clinical pathway for women presenting with SUI with or without pelvic prolapse.

Surgical method Patients participating in this study will undergo standard preoperative and peri-operative care, and anesthetic and pain management care, identical than that which occurs for any pelvic reconstructive surgery within our division. Coexisting pelvic prolapse repairs such as cystocele and rectocele repair, with or without hysterectomy, will be performed per routine.

For treating SUI, the dissection will be completely identical to mid-urethral sling. The difference will be instead of passing the mesh through the tunnels on each side of urethra and exiting through rectus fascia, the investigators will use a ¾ x ⅜ inch polypropylene mesh and place it under the mid urethral. This mesh will be suspended by two suspending permanent sutures on each side to the pubic rami periosteum. At this point sutures will be tied down and the vaginal skin closed with a 2-0 vicryl suture.

Postoperative care This procedure entails no additional or specific post-operative activity limitations or care in comparison to the existing baseline pelvic organ prolapse surgeries. The investigators anticipate that all patients will be discharged from the hospital consistent with normal patterns, either on the same day of surgery or after a brief hospital stay, depending on the meeting of postoperative milestones and discharge criteria.

Follow up Patients will return to the office for postoperative visits at 2 weeks, 2 months, and 12 months after surgery. During the 2-month and 12 month follow-up visits, a vaginal exam and pelvic floor ultrasound will be performed to evaluate healing and urethral motion.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic stress urinary incontinence

Exclusion Criteria:

* Women of childbearing age (0-45 years)
* Previous stress urinary incontinence surgery

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Stress urinary incontinence in women.
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFDI-20 score | 12 months post-op
  Pelvic Floor Disability Index (PFDI-20) score indicating SUI symptom severity. Higher values indicate greater distress or worse outcome. The sub-scales score ranges from 0 to 100. The summary score ranges from 0 to 300.

SECONDARY OUTCOMES:
Complication measured by distal urethral swing angle | 12 months post-op
  Investigate the efficacy of this mesh-reduced suture based surgical technique on key urethral support defects observed with 3D ultrasound.
  This will be measured by distal urethral swing angle during Valsalva measured via pelvic ultrasound.
Complication measured by proximal urethral swing angle | 12 months post-op
  Investigate the efficacy of this mesh-reduced suture based surgical technique on key urethral support defects observed with 3D ultrasound.
  This will be measured by proximal urethral swing angle during Valsalva measured via pelvic ultrasound.
Complication measured by early and remote post-operative complications | 12 months post-op
  Investigate the efficacy of this mesh-reduced suture based surgical technique on key urethral support defects observed with 3D ultrasound.
  This will be measured by early and remote postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Chill, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University Health System, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with other investigators listed in the study within NorthShore University Health System.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available during data collection until after publication.
Access Criteria: Other investigators within NorthShore University Health System who are listed on the study delegation log will receive individual participant data during data collection for use during data analysis.

REFERENCES:
- [Background] Ford AA, Rogerson L, Cody JD, Ogah J. Mid-urethral sling operations for stress urinary incontinence in women. Cochrane Database Syst Rev. 2015 Jul 1;(7):CD006375. doi: 10.1002/14651858.CD006375.pub3. PMID 26130017
- [Background] Richter HE, Albo ME, Zyczynski HM, Kenton K, Norton PA, Sirls LT, Kraus SR, Chai TC, Lemack GE, Dandreo KJ, Varner RE, Menefee S, Ghetti C, Brubaker L, Nygaard I, Khandwala S, Rozanski TA, Johnson H, Schaffer J, Stoddard AM, Holley RL, Nager CW, Moalli P, Mueller E, Arisco AM, Corton M, Tennstedt S, Chang TD, Gormley EA, Litman HJ; Urinary Incontinence Treatment Network. Retropubic versus transobturator midurethral slings for stress incontinence. N Engl J Med. 2010 Jun 3;362(22):2066-76. doi: 10.1056/NEJMoa0912658. Epub 2010 May 17. PMID 20479459
- [Background] Kenton K, Stoddard AM, Zyczynski H, Albo M, Rickey L, Norton P, Wai C, Kraus SR, Sirls LT, Kusek JW, Litman HJ, Chang RP, Richter HE. 5-year longitudinal followup after retropubic and transobturator mid urethral slings. J Urol. 2015 Jan;193(1):203-10. doi: 10.1016/j.juro.2014.08.089. Epub 2014 Aug 23. PMID 25158274
- [Background] Nolfi AL, Brown BN, Liang R, Palcsey SL, Bonidie MJ, Abramowitch SD, Moalli PA. Host response to synthetic mesh in women with mesh complications. Am J Obstet Gynecol. 2016 Aug;215(2):206.e1-8. doi: 10.1016/j.ajog.2016.04.008. Epub 2016 Apr 16. PMID 27094962
- [Background] Frenkl TL, Rackley RR, Vasavada SP, Goldman HB. Management of iatrogenic foreign bodies of the bladder and urethra following pelvic floor surgery. Neurourol Urodyn. 2008;27(6):491-5. doi: 10.1002/nau.20558. PMID 18537142
- [Background] Brubaker L, Norton PA, Albo ME, Chai TC, Dandreo KJ, Lloyd KL, Lowder JL, Sirls LT, Lemack GE, Arisco AM, Xu Y, Kusek JW; Urinary Incontinence Treatment Network. Adverse events over two years after retropubic or transobturator midurethral sling surgery: findings from the Trial of Midurethral Slings (TOMUS) study. Am J Obstet Gynecol. 2011 Nov;205(5):498.e1-6. doi: 10.1016/j.ajog.2011.07.011. Epub 2011 Jul 20. PMID 21925636
- [Background] Baracat F, Mitre AI, Kanashiro H, Montellato NI. Endoscopic treatment of vesical and urethral perforations after tension-free vaginal tape (TVT) procedure for female stress urinary incontinence. Clinics (Sao Paulo). 2005 Oct;60(5):397-400. doi: 10.1590/s1807-59322005000500008. Epub 2005 Oct 24. PMID 16254676
- [Background] Giri SK, Drumm J, Flood HD. Endoscopic holmium laser excision of intravesical tension-free vaginal tape and polypropylene suture after anti-incontinence procedures. J Urol. 2005 Oct;174(4 Pt 1):1306-7. doi: 10.1097/01.ju.0000173926.04596.55. PMID 16145408
- [Background] Molden SM, Lucente VR. New minimally invasive slings: TVT Secur. Curr Urol Rep. 2008 Sep;9(5):358-61. doi: 10.1007/s11934-008-0062-8. PMID 18702918
- [Background] Palma P, Riccetto C, Bronzatto E, Castro R, Altuna S. What is the best indication for single-incision Ophira Mini Sling? Insights from a 2-year follow-up international multicentric study. Int Urogynecol J. 2014 May;25(5):637-43. doi: 10.1007/s00192-013-2242-4. Epub 2013 Oct 30. PMID 24170223
- [Background] Talley NJ, Weaver AL, Zinsmeister AR, Melton LJ 3rd. Functional constipation and outlet delay: a population-based study. Gastroenterology. 1993 Sep;105(3):781-90. doi: 10.1016/0016-5085(93)90896-k. PMID 8359649
- [Background] Talley NJ, Fleming KC, Evans JM, O'Keefe EA, Weaver AL, Zinsmeister AR, Melton LJ 3rd. Constipation in an elderly community: a study of prevalence and potential risk factors. Am J Gastroenterol. 1996 Jan;91(1):19-25. PMID 8561137
- [Background] Riss S, Stift A. Surgery for obstructed defecation syndrome - is there an ideal technique. World J Gastroenterol. 2015 Jan 7;21(1):1-5. doi: 10.3748/wjg.v21.i1.1. PMID 25574075
- [Background] Bordeianou L, Paquette I, Johnson E, Holubar SD, Gaertner W, Feingold DL, Steele SR. Clinical Practice Guidelines for the Treatment of Rectal Prolapse. Dis Colon Rectum. 2017 Nov;60(11):1121-1131. doi: 10.1097/DCR.0000000000000889. No abstract available. PMID 28991074